CLINICAL TRIAL: NCT01110044
Title: Immunogenicity and Safety of a Birth Dose of GlaxoSmithKline Biologicals' Reduced-antigen-content Tri-component Pertussis (251154) Vaccine
Brief Title: Study of a Birth Dose of GlaxoSmithKline Biologicals' 251154 Vaccine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was cancelled before enrolment for reasons not related to vaccine safety or efficacy.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112980
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Infections, Rotavirus
Keywords: Neonatal vaccination
MeSH Terms: conditions — Rotavirus Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; PHiD-CV vaccine; RIX4414 vaccine

ARMS (2):
- Group A (Experimental): Subjects will be administered 251154 vaccine at birth, Infanrix hexa™ at 2, 4, 6 and 12-18 months of age, Synflorix™ at 2, 4, 6 and 12-18 months of age, Rotarix™ at 2 and 4 months of age.
  Interventions: Biological: 251154 vaccine; Biological: Infanrix hexa™; Biological: Synflorix™; Biological: Rotarix™
- Group B (Active Comparator): Subjects will be administered no vaccine at birth, Infanrix hexa™ at 2, 4, 6 and 12-18 months of age, Synflorix™ at 2, 4, 6 and 12-18 months of age, Rotarix™ at 2 and 4 months of age.
  Interventions: Biological: Infanrix hexa™; Biological: Synflorix™; Biological: Rotarix™

INTERVENTIONS:
Biological: 251154 vaccine — Intramuscular, single dose
  Arms: Group A
Biological: Infanrix hexa™ — Intramuscular, four doses
Biological: Synflorix™ — Intramuscular, four doses
Biological: Rotarix™ — Oral, two doses

SUMMARY:
The purpose of the study is to evaluate the safety and immunogenicity of a birth dose of GSK Biologicals' reduced-antigen-content tri-component pertussis (251154) vaccine followed by routine paediatric vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/LAR(s) can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* A male or female infant between, and including, 2 and 5 days of age at the time of randomisation.
* Subjects who are born after an uncomplicated gestation period of 36 to 42 weeks inclusive.
* Subjects born to a mother seronegative for hepatitis B surface antigen.
* Subjects with a birth weight >= 2.5 kg.
* Subjects with a 5-minute Apgar score >= 7.
* Healthy subjects as established by medical history and clinical examination

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines since birth, or planned use during the study period.
* Born to a mother known or suspected to be seropositive for HIV.
* Family history of congenital or hereditary immunodeficiency.
* Children in care..
* Neonatal jaundice requiring systemic treatment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of any vaccine since birth or planned administration during the study period with the exception of inactivated influenza vaccines.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* History of seizures or progressive neurological disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Major congenital defects or serious chronic illness, including perinatal brain damage.

The following condition is temporary or self-limiting, and a subject may be vaccinated once the condition has resolved if no other exclusion criteria is met:

• Current febrile illness or temperature >= 38.5°C on oral or axillary setting, or >= 39.0°C on rectal setting, or other moderate to severe illness within 24 hours of study vaccine administration.

Ages: 2 Days to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity with respect to components of the study vaccines. | One month after the first dose of primary vaccination.
Immunogenicity with respect to components of the study vaccines. | One month after the third dose of primary vaccination.

SECONDARY OUTCOMES:
Immunogenicity with respect to components of the study vaccines (on secondary readouts). | One month after the second dose of primary vaccination.
Immunogenicity with respect to components of the study vaccines (on secondary readouts). | One month after the third dose of primary vaccination.
Immunogenicity with respect to components of the study vaccines (on secondary readouts). | One month after booster vaccination.
Occurrence of solicited local and general symptoms (on secondary readouts). | On Day 0-Day 7 after neonatal vaccination.
Occurrence of solicited local and general symptoms (on secondary readouts). | On Day 0-Day 3 after each dose of primary and booster vaccination.
Occurrence of unsolicited adverse events (on secondary readouts). | On Day 0-Day 30 after each vaccination.
Occurrence of serious adverse events (on secondary readouts). | From enrolment up to study end.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline